CLINICAL TRIAL: NCT01770119
Title: Induction and Maintenance of Immunity Against Measles in Pediatric Orthotopic Liver Transplantation Recipients: a Prospective Nationwide Study in Switzerland
Brief Title: Induction of Immunity Against Measles in Pediatric Liver Transplant Recipients
Acronym: MMRinOLT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Klara M. Pósfay Barbe (Other)
Collaborators: University Hospital, Geneva (Other)
Responsible Party: Sponsor-Investigator, Klara M. Pósfay Barbe, Head of Pediatric Infectious Diseases, University Hospital, Geneva
Organization: University Hospital, Geneva (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MMR in pediatric OLT; 12-226 (MatPed 12-048) (Other: IRB)
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Measles
Keywords: Measles; Mumps; Rubella; Pediatric; Solid-organ transplant; serology; vaccine
MeSH Terms: conditions — Measles; Mumps; Rubella

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MMR vaccination (Experimental): MMR vaccine to seronegative pediatric SOT recipients
  Interventions: Biological: MMR vaccination

INTERVENTIONS:
Biological: MMR vaccination — Unprotected children will be vaccinated with two MMR vaccines

SUMMARY:
Measles is a vaccine-preventable disease, which can be life-threatening in immunosuppressed children. Currently, measles vaccine is not recommended in pediatric orthotopic liver transplant recipients, because it is a live-attenuated vaccine.

We want to assess the influence of immunosuppression on immunity against measles in previously vaccinated children and to evaluate the induction of B cell and T cell response against measles elicited by vaccination in children at least 12 months after transplantation.

DETAILED DESCRIPTION:
Eligible children in Group 2 will receive a standard dose (0.5 ml) of MMR vaccine during the first medical visit (V1). The lot number and the expiration date will both be recorded on the patient's case report form (CRF). A serological evaluation 4-8 weeks after MMR will identify children requiring an additional dose given 1-2 months apart, as currently recommended for subjects 1 year-old or with limited immune competence (i.e. HIV-infected children). Serological evaluation 4-8 weeks after the second dose or at the one-year follow-up will identify eventual non-responder requiring a third dose. Three will be the maximal number of administrated dose according to this protocol. The persistence of measles-specific antibodies will be assessed yearly, when patients come for their routine visit to the transplant center.

Children who do not need MMR immunization because of protective levels will be monitored yearly for maintenance of antibody levels during routine yearly visits/ blood samplings and will not have further intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 12 months
* Measles-specific IgG antibodies negative (<0.2 IU/L), as detected by the routine ELISA assay
* ≥ 12 months from the time of transplantation and ≥ 2 months from the time of an acute rejection episode
* Steroids < 2 mg/kg/day, tacrolimus < 0.3mg/kg/day and tacrolimus level < 8 ng/ml for > 1 month.
* Total lymphocyte count ≥ 750 cells/ul at time of immunization

Exclusion Criteria:

* Known wild-type measles exposure during the last four weeks
* Measles-containing immunoglobulins administered within the 5 months preceding the measles vaccine. If the child receives measles-containing Ig before an additional dose of MMR vaccine, he/she will be withdrawn from the study
* Antiviral agents administered during the last four weeks
* Febrile illness (>38.5°) in the 72 hours before vaccine administration
* Chronic aspirin therapy
* Any other immunization with a live-attenuated vaccine during the last four weeks
* Pregnancy

Ages: 12 Months to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2013-04; Primary Completion 2022-04 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
serologic response to MMR vaccine in seronegative transplant recipients | 2 months after vaccination
  Pediatric transplant recipients will be vaccinated with MMR vaccine (previously seronegative) and their seroresponse will be measured 2 months later

SECONDARY OUTCOMES:
Persistance of seroresponse to MMR vaccine | 3 years
  Seroresponse to MMR vaccine will be followed over time in pediatric transplant recipients

OTHER OUTCOMES:
Efficacy of MMR vaccine in pediatric SOT recipients | 3 years
  Protection against vaccine-preventable diseases will be assessed in pediatric SOT recipients

CONTACTS AND LOCATIONS:
Overall Officials: Klara M Posfay-Barbe, MD, MS, Principal Investigator — University Hospitals of Geneva
Locations (1):
- Children's Hospital of Geneva, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pittet LF, Verolet CM, McLin VA, Wildhaber BE, Rodriguez M, Cherpillod P, Kaiser L, Siegrist CA, Posfay-Barbe KM. Multimodal safety assessment of measles-mumps-rubella vaccination after pediatric liver transplantation. Am J Transplant. 2019 Mar;19(3):844-854. doi: 10.1111/ajt.15101. Epub 2018 Oct 1. PMID 30171797
- [Background] Suresh S, Upton J, Green M, Pham-Huy A, Posfay-Barbe KM, Michaels MG, Top KA, Avitzur Y, Burton C, Chong PP, Danziger-Isakov L, Dipchand AI, Hebert D, Kumar D, Morris SK, Nalli N, Ng VL, Nicholas SK, Robinson JL, Solomon M, Tapiero B, Verma A, Walter JE, Allen UD. Live vaccines after pediatric solid organ transplant: Proceedings of a consensus meeting, 2018. Pediatr Transplant. 2019 Nov;23(7):e13571. doi: 10.1111/petr.13571. Epub 2019 Sep 9. PMID 31497926